CLINICAL TRIAL: NCT03044444
Title: Establishing the Effect of Long-term Citrus Extract Supplementation on Exercise-specific Performance in Moderately Trained Athletes
Brief Title: The Effect of a Citrus Extract on Exercise Performance in Moderately Trained Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioActor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HES_PER_002
Record Dates: First submitted 2017-01-30; First posted 2017-02-07 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Exercise Performance
Keywords: performance; polyphenols; nutrition; sports
MeSH Terms: interventions — grapefruit seed extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high dose citrus extract (Experimental): this group will receive a high dose (500mg/day) of the citrus extract for 8 weeks
  Interventions: Dietary Supplement: citrus extract
- low dose citrus extract (Experimental): this group will receive a low dose (400mg/day) of the citrus extract for 8 weeks
  Interventions: Dietary Supplement: citrus extract
- placebo (Placebo Comparator): this group will receive a placebo (500mg maltodextrin per day) for 8 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: citrus extract — Participants will receive either a low or high dose citrus extract
  Arms: high dose citrus extract; low dose citrus extract
Other: placebo — participants will receive 500mg of maltodextrin
  Arms: placebo

SUMMARY:
In this study, the effect of citrus extract on exercise performance will be investigated. The study consists of three groups: one group will receive a high dose citrus extract, one group will receive a low dose citrus extract and the last group will receive a placebo. After four and eight weeks the effects on performance are measured through a Wingate cycling test. It is expected that exercise performance will increase in the citrus extract groups, compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* healthy idividuals
* Participants are amateur or (semi-) professional athletes in resistance or interval sports (engage in >4 hours of intense physical activity per week).

Exclusion Criteria:

* Use of creatine supplements and/or anabolic steroids.
* Allergy to test product/placebo
* Allergy to citrus fruits
* BMI lower than 18 or higher than 30
* Recent muscle injury in less than one month before the start of the study.
* Cardiovascular complications
* Use of medication that may interfere with the study results
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study.
* Abuse of products; alcohol (> 20 alcoholic units per week) and drugs.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
peak force output Wingate | 8 weeks
  Peak force output in Watts during a high intensity repeated sprint cycling exercise

SECONDARY OUTCOMES:
jumping height | 8 weeks
  jumping height in cm measured during a vertical jump exercise
peak force output Handgrip | 8 weeks
  Peak force output in Watts during a handgrip strength test
force output Jump | 8 weeks
  force output in W measured during a vertical jump exercise
anaerobic capacity | 8 weeks
  total amount of power (W) generated in the first 30 seconds of the the triple Wingate cycle test
running time | 8 weeks
  running time in minutes and seconds measured over 1600m

OTHER OUTCOMES:
lactate | 8 weeks
  post-exercise blood lactate in mmol/L after triple Wingate cycle exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Troost, Dr., Principal Investigator — Maastricht University
Locations (1):
- High Performance Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Iersel LE, Stevens YR, Conchillo JM, Troost FJ. The effect of citrus flavonoid extract supplementation on anaerobic capacity in moderately trained athletes: a randomized controlled trial. J Int Soc Sports Nutr. 2021 Jan 6;18(1):2. doi: 10.1186/s12970-020-00399-w. PMID 33407631